CLINICAL TRIAL: NCT05326724
Title: The Role of Acupuncture-induced Exosome in Treating Post-stroke Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH111-REC2-024
Record Dates: First submitted 2022-03-28; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Exosome; Post-stroke Dementia; Acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture (Experimental)
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — The stainless steel needles are used to insert into the three points of Sishencong and the Baihui, and the Dazhui, once a week, once for 20 minutes, for 12 consecutive weeks.

SUMMARY:
Stroke is the main cause of disability and the second main cause of dementia. Approximately 21.5% of patients develop dementia within 4 years after stroke. The main clinical manifestation of dementia is memory and cognitive impairment. At present, acetylcholinesterase inhibitors and NMDA glutamate receptor antagonists, were used for dementia treatment, but those drugs have limited efficacy. Exosome is an extracellular vesicle from the endosomal, size range from ~40 to 160 nm (average ~100 nm). It contains many cells including DNA, RNA, fat, and metabolites, as well as cytoplasm and cell surface proteins that play a role in regulating intercellular communication. Some studies believe that exosomes in the circulation are an ideal marker to reflect the pathological progress and recovery of stroke, and play a key role in the reorganization of tissues and the progress of neurodegeneration after stroke. Our previous studies have known that acupuncture can increase the long-term potentiation of hippocampal CA1 in rats with ischemic stroke, and improve learning-memory and neurological function. Therefore, the purpose of this study is to explore the role of acupuncture-induced exosome in the treatment of post-stroke dementia.

ELIGIBILITY:
Inclusion Criteria:

1. History of stroke.
2. MMSE score between 16 and 26.

Exclusion Criteria:

1. Those with serious diseases, such as heart failure, chronic failure or cancer patients, etc.
2. Intolerance to acupuncture treatment.
3. Allergy to acupuncture needles.
4. Refusal to sign the informed consent form.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
concentration of Exosome | 12 weeks
Alzheimer's Disease Assessment Scale-Cognitive Subscale scale | 12 weeks
  Higher scores indicate greater cognitive impairment.
Behavioural and Psychological Symptoms of Dementia scale | 12 weeks
  The greater cognitive impairment or dementia severity is associated with higher rates of some BPSD (Behavioral and psychological symptoms of dementia ).

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan